CLINICAL TRIAL: NCT00329160
Title: A Study to Evaluate the Efficacy and Safety of Rosuvastatin in the Long-term Treatment of Hypercholesterolaemic Subjects With Coronary Heart Disease as Measured by Intravascular Ultrasonography
Brief Title: Rosuvastatin in the Long-term Treatment of Hypercholesterolaemic Subjects With Coronary Heart Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Shionogi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D3565L00002; 0407E1841
Record Dates: First submitted 2006-05-22; First posted 2006-05-24 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2011-08

CONDITIONS: Hypercholesteremia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Rosuvastatin Calcium; Hydroxymethylglutaryl-CoA Reductase Inhibitors

INTERVENTIONS:
Drug: Rosuvastatin — 2.5-20 mg
Drug: HMG CoA inhibitor — 3-hydroxy-3-methylglutaryl-coenzyme A

SUMMARY:
The primary objective of this study is to evaluate that 76 weeks of treatment with rosuvastatin calcium 2.5-20 mg results in no progression of coronary artery atherosclerotic volume as measured by intravascular ultrasonography (IVUS) imaging in hypercholesterolaemic subjects with coronary heart disease (CHD).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent,
* 20 to 75 years old,
* Plan to undergo coronary angiography (CAG) or Percutaneous coronary intervention (PCI) and LDL-C ≥ 140 mg/dL (untreated patients) or LDL-C ≥ 100 mg/dL (treated patients)

Exclusion Criteria:

* Acute myocardial infarction within 72 hours after the onset,
* Heart failure of New York Heart Association (NYHA) Class III or above,
* Serious arrhythmia,
* Being treated with LDL-apheresis
* History of serious reaction or hypersensitivity to other HMG-CoA reductase inhibitors.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2005-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masunori Matsuzaki, MD, Principal Investigator — Yamaguchi University Hospital
Locations (27):
- Japan (27):
  - Research Site, Gifu
  - Research Site, Hamada
  - Research Site, Hiroshima
  - Research Site, Ichinomiya
  - Research Site, Inba-mura
  - Research Site, Izumi
  - Research Site, Izumisano
  - Research Site, Izumo
  - Research Site, Kagoshima
  - Research Site, Kanazawa
  - Research Site, Kasuga
  - Research Site, Kobe
  - Research Site, Komaki
  - Research Site, Konancho
  - Research Site, Kumamoto
  - Research Site, Kurume
  - Research Site, Kyoto
  - Research Site, Osaka
  - Research Site, Ōmiya
  - Research Site, Sapporo
  - Research Site, Shinjō
  - Research Site, Shūnan
  - Research Site, Suita
  - Research Site, Tokyo
  - Research Site, Ube
  - Research Site, Yamaguchi
  - Research Site, Yokohama

REFERENCES:
- [Derived] Daida H, Takayama T, Hiro T, Yamagishi M, Hirayama A, Saito S, Yamaguchi T, Matsuzaki M; COSMOS Investigators. High HbA1c levels correlate with reduced plaque regression during statin treatment in patients with stable coronary artery disease: results of the coronary atherosclerosis study measuring effects of rosuvastatin using intravascular ultrasound in Japanese subjects (COSMOS). Cardiovasc Diabetol. 2012 Jul 25;11:87. doi: 10.1186/1475-2840-11-87. PMID 22831708

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Observation Period :Prior to study-related activities, all subjects will sign an informed consent form. IVUS and CAG is performed prior Treatment Treatment Period: Eligible patients started treatment; rosuvastatin 2.5 mg once daily; those whose LDL-C remained >80 mg/dl after 4 wks of treatment, the dose can be titrated to a maximum of 20 mg/day
Groups:
- Rosuvastatin: rosuvastatin 2.5 mg once daily; in those whose LDL-C remained >80 mg/dl after 4 weeks of treatment, the dosage could be titrated up to a maximum of 20 mg/day, which is the highest approved regimen by the Ministry of Health, Labor and Welfare of Japan. Subjects attended follow-up visits every 4 weeks over 76 weeks after starting treatment with rosuvastatin.
Period: Overall Study
Arm/Group | Rosuvastatin
Started | 214
Observation Period | 214
Treatment Period | 214
Completed | 126
Not Completed | 88
Not completed — Adverse Event | 27
Not completed — Withdrawal by Subject | 13
Not completed — Protocol Violation | 2
Not completed — Did not Receive Study Drug | 1
Not completed — Incomplete IVUS | 45

BASELINE CHARACTERISTICS:
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 126
Age Continuous [Mean (Standard Deviation); unit: years]
  Years | 62.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants] — 1 participant did not receive drug and is not captured in these figures
  Participants
    Female | 30
    Male | 96

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline (Before the Start of Rosuvastatin Treatment) to Week 76 in the Plaque Volume (PV)
Description: Plaque volume will be assessed by volumetric analysis with the echoPlaque2 system (Indec Systems Inc). Baseline and follow-up IVUS images will be reviewed side-by-side on a display, and the target segment selected. The target segment to be monitored will be determined in a non-PCI site (>5 mm proximal or distal to the PCI site) with a reproducible index such as side branches, calcifications, or stent edges.
Time Frame: Baseline and 76 weeks
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 126
Percent Change | 14.1 (-5.066)

2. Secondary Outcome: Change From Baseline to Week 76 in Plaque Volume (PV) in the Target Lesion
Description: Target Lesion indicates Coronary plaque composition of culprit lesions.
Time Frame: Baseline - 76Weeks
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 126
mg/dL | 12.074 (-5.259)

3. Secondary Outcome: Percent Change From Baseline to Specified Measurement Time Points in Low-density Lipoprotein （LDL-C）
Time Frame: Baseline - 76Weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 126
Percent change | 16.9 (-38.6)

4. Secondary Outcome: Percent Change in High-sensitivity C-reactive Protein (HS-CRP) From Baseline to Specified Measurement Time Points
Time Frame: Baseline - 76Weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Rosuvastatin
Number analyzed (Participants) | 126
Percent change | 18.1 (291.3)

ADVERSE EVENTS:
Arm/Group | Rosuvastatin
Serious Adverse Events (participants affected / at risk) | 98/213
Other Adverse Events (participants affected / at risk) | 588/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin (N=213)
Anaemia (Blood and lymphatic system disorders) | 1
Acute Myocardial Infarction (Cardiac disorders) | 1
Angina Pectoris (Cardiac disorders) | 7
Angina Unstable (Cardiac disorders) | 1
Atrioventricular Block (Cardiac disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Cardiac Failure Acute (Cardiac disorders) | 1
Cardiac Failure Congestive (Cardiac disorders) | 2
Coronary Artery Perforation (Cardiac disorders) | 1
Coronary Artery Stenosis (Cardiac disorders) | 21
Prinzmetal Angina (Cardiac disorders) | 2
Cataract (Eye disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Rectal Ulcer (Gastrointestinal disorders) | 1
Oedema Peripheral (General disorders) | 1
Puncture Site Haemorrhage (General disorders) | 1
Pyrexia (General disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 2
Liver Disorder (Hepatobiliary disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Filariasis (Infections and infestations) | 1
Liver Abscess (Infections and infestations) | 1
Brain Contusion (Injury, poisoning and procedural complications) | 1
Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 2
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1
In-Stent Coronary Artery Restenosis (Injury, poisoning and procedural complications) | 2
Stent Occlusion (Injury, poisoning and procedural complications) | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 2
Alanine Aminotransferase Increased (Injury, poisoning and procedural complications) | 1
Aspartate Aminotransferase Increased (Injury, poisoning and procedural complications) | 1
Blood Alkaline Phosphatase Increased (Injury, poisoning and procedural complications) | 1
Blood Bilirubin Increased (Injury, poisoning and procedural complications) | 1
Blood Pressure Decreased (Injury, poisoning and procedural complications) | 1
C-Reactive Protein Increased (Injury, poisoning and procedural complications) | 2
Gamma-Glutamyltransferase Increased (Injury, poisoning and procedural complications) | 1
Glycosylated Haemoglobin Increased (Injury, poisoning and procedural complications) | 1
Neutrophil Count Decreased (Injury, poisoning and procedural complications) | 1
Platelet Count Decreased (Injury, poisoning and procedural complications) | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Large Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Small Cell Lung Cancer Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral Haemorrhage (Nervous system disorders) | 1
Cerebral Infarction (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Facial Palsy (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Loss Of Consciousness (Nervous system disorders) | 1
Thalamus Haemorrhage (Nervous system disorders) | 1
Visual Field Defect (Nervous system disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Haemorrhage Subcutaneous (Skin and subcutaneous tissue disorders) | 1
Arterial Bypass Operation (Surgical and medical procedures) | 1
Coronary Angioplasty (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rosuvastatin (N=214)
Constipation (Gastrointestinal disorders) | 14
Dental Caries (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 12
Nasopharyngitis (Infections and infestations) | 69
Alanine Aminotransferase Increased (Infections and infestations) | 38
Aspartate Aminotransferase Increased (Infections and infestations) | 28
Blood Alkaline Phosphatase Increased (Infections and infestations) | 20
Blood Creatine Phosphokinase Increased (Infections and infestations) | 43
Blood Pressure Increased (Infections and infestations) | 22
Blood Urine Present (Infections and infestations) | 33
C-Reactive Protein Increased (Infections and infestations) | 16
Gamma-Glutamyltransferase Increased (Infections and infestations) | 48
Glucose Urine Present (Infections and infestations) | 28
Glycosylated Haemoglobin Increased (Infections and infestations) | 12
Haematocrit Decreased (Infections and infestations) | 12
Haemoglobin Decreased (Infections and infestations) | 14
Protein Urine Present (Infections and infestations) | 31
Red Blood Cell Count Decreased (Infections and infestations) | 11
White Blood Cell Count Increased (Infections and infestations) | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 11
Dizziness (Nervous system disorders) | 19
Headache (Nervous system disorders) | 11
Insomnia (Psychiatric disorders) | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 18

LIMITATIONS AND CAVEATS:
Because there was no placebo arm the net effect of rosuvastatin was not clarified. This study examined only single measurable plaques, which might not represent pan-coronary nature of plaque.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other